CLINICAL TRIAL: NCT03178058
Title: Risk Factors for Nausea, Vomiting and Pruritus After Neuraxial Morphine for Cesarean Section
Brief Title: Risk Factors for Postoperative Nausea, Vomiting and Pruritus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharon orbach, Dr, Rabin Medical Center
Other Study IDs: 0387-15
Record Dates: First submitted 2017-05-09; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parturients for CS: Parturients presenting for Cesarean section will be enrolled preoperatively. Prior to surgery women will be given a questionnaire detailing previous motion sickness, previous history of PONV, emesis during pregnancy, smoking history , itching history, skin atopy and allergies. After surgery details about surgery will be added: intraoperative hypotension, use of phenylepherine, intraoperative nausea and vomiting, exteriorization of uterus, extent of adhesions, need for uterotonic medications, and estimated bleeding.
  Parturients will be assessed 1 hour and 24 postoperatively by attending anesthesiologist, PONV incidence will be reported using a three point ordinal scale (0 = none, 1 = nausea, 2 = retching, 3 =vomiting).
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — Prior to surgery women will be given a questionnaire detailing previous motion sickness, previous history of PONV, emesis during pregnancy, smoking history , itching history, skin atopy and allergies. After surgery details about surgery will be added: intraoperative hypotension, use of phenylepherine, intraoperative nausea and vomiting, exteriorization of uterus, extent of adhesions, need for uterotonic medications, and estimated bleeding.
  Parturients will be assessed 1 hour and 24 postoperatively by attending anesthesiologist, PONV incidence will be reported using a three point ordinal scale (0 = none, 1 = nausea, 2 = retching, 3 =vomiting).

SUMMARY:
In this study we would like to identify demographic and individual risk factors that place parturients at a higher risk for postoperative nausea and vomiting (PONV) and itching following administered neuraxial morphine for cesarean section. Our primary objective is to develop a reliable predictive neuraxial morphine induced nausea and vomiting (NMINV) and itching model.

DETAILED DESCRIPTION:
Introduction Neuraxial morphine provides effective and long-lasting analgesia after cesarean section. It is currently considered the gold standard for postoperative pain. However, it is associated with problematic side effects including nausea and vomiting, pruritus, and rarely respiratory depression.

Postoperative nausea and vomiting (PONV) occurs in up to 60-80% of parturients receiving neuraxial opioid administration , and reported incidence of pruritus varies from 30% to 100%.

A wide range of pharmaceutical and non pharmaceutical agents are commonly used in clinical practice for the treatment and prophylaxis of neuraxial morphine induced postoperative nausea, vomiting and pruritus. Antiemetic medications such as droperidol, dexamethasone, metoclopramide and ondansetron, have been studied for their efficacy in preventing PONV . Despite the wide variety of these available drugs, many of them are ineffective and have side effects. Dexamethasone ,for example, although it has been proven as an effective antiemetic in patients receiving epidural morphine, it is ineffective monotherapy in patients receiving intrathecal morphine . In addition it is associated severe perineal pruritus . Common side effects of ondansetron are headache, flushing, dizziness and constipation. Droperidol is associated with undesirable side effects: sedation, hypotension, and extrapy-ramidal reactions . Both droperidol and ondansetron are known to prolong the QTc interval.

To date although pruritus after neuraxial administration of morphine is a common side effect, there is little available effective treatment . Studies have found opioid-induced pruritus to be dose dependent and minimal analgesic doses of opioids are recommended. Several agents from numerous drug families have been employed, although none has proved to be totally effective . Treatment medications include: naloxone, nalbuphine, diphenhydramine and droperidol .

To date there are no studies which have identified risk factors for PONV and pruritus after administration of nauraxial morphine. Attempts have been made to identify which patients are at risk for PONV after general anesthesia .

There are anesthetic, surgical, and individual risk factors are linked to PONV Studies in this field have identified several predicting risk factors for PONV .

Apfel et al established a validated simplified scoring systems to assess risk factors for nausea and vomiting after general anesthesia. His simplified sum score system included four risk factors: female gender, prior history of motion sickness or PONV, nonsmoking, and the use of postoperative opioids .

If none or only one risk factor is present the predicted incidence of PONV may vary between about 10% and 21%, whereas if at least two risk factors are present it increases to between 39% and 78%.

To date research has yet to yield a predictive model for neuraxial morphine induced nausea and vomiting (NMINV). Likewise risk factor for neuraxial itching have yet to be established.

Methods This is a prospective, single center study, which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital. The Institutional Review Board has approved this study.

All women undergoing cesarean section delivery under spinal anesthesia with neuraxial morphine will be enrolled after filling out an informed consent prior to surgery. Women undergo spinal anesthesia with 10-12 mg heavy bupivicaine, 20 ucg fentanyl and 100 ucg morphine. Phenylepherine drip is used at anesthesiologist's discretion. If not treatment dose of ephedrine or phenylepherine are given as required by blood pressure.

All women receive prophylaxis intravenous dexamenthasone 4 mg and prophylactic intravenous ondansetron 4mg, as standard departmental protocol.

Prior to surgery women will be given a questionnaire detailing previous motion sickness, previous history of PONV, emesis during pregnancy, smoking history , itching history, skin atopy and allergies. After surgery details about surgery will be added: intraoperative hypotension, use of phenylepherine, intraoperative nausea and vomiting, exteriorization of uterus, extent of adhesions, need for uterotonic medications, and estimated bleeding.

Parturients will be assessed 1 hour and 24 postoperatively by attending anesthesiologist, PONV incidence will be reported using a three point ordinal scale (0 = none, 1 = nausea, 2 = retching, 3 =vomiting).

Nausea includes any feeling of sickness with an inclination to vomit. Retching includes any reverse movement of the stomach and esophagus without vomiting, including attempting vomiting.

Vomiting is defined as the involuntary, forceful expulsion of one's gastric contents through the mouth and sometimes the nose.

A VNRS (vas numerical rating score) (from 0-10 0= no itching at all , 10= worst itching possible) will be used to measure overall presence and severity of pruritus.

Any severe incidence of VNRS defined above 7 will be noted. All parturients need for postoperative antiemetic and antipruritic medications will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 undergoing cesarean section under spinal anesthesia with intrathecal morphine in Beilinson Hospital following obtaining written informed consents forums with the ability to comply with the study requirements will be included in our study.

Exclusion Criteria:

* Women under age 18, women undergoing cesarean section under general anesthesia or under spinal anesthesia without intrathecal morphine and women who don't understand the inform consent form will be excluded from participating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort consists of parturients presenting for cesarean section under spinal anesthesia with intrathecal morphine above the age 18.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Demographic causative factors for postoperative nausea after administration of neuraxial morphine | 24 Hours
  Demographic factors that contribute to postoperative nausea after administration of neuraxial morphine as measured by the PONV questionnaire

SECONDARY OUTCOMES:
Demographic causative factors for postoperative vomiting after administration of neuraxial morphine | 24 hours
  emographic factors that contribute to postoperative vomiting after administration of neuraxial morphine as measured by the PONV questionnaire
Demographic causative factors for postoperative pruritus after administration of neuraxial morphine | 24 hours
  Demographic factors that contribute to postoperative pruritus after administration of neuraxial morphine as measured by the PONV questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel